CLINICAL TRIAL: NCT05372263
Title: Safety Surveillance of Targeted Drugs for Pulmonary Hypertension Using a Computerized Follow-up System: a Nationwide Cohort Study
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lu Hua, Chief Physician, China National Center for Cardiovascular Diseases
Other Study IDs: CST2020CT303
Record Dates: First submitted 2022-04-28; First posted 2022-05-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recruit at least 700 PH patients, follow up every 6 months based on a computerized follow-up system. Primary outcomes are adverse drug events and all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Age from 3 months to 85 years, no sex preference;
* Right heart catheter meet the following conditions simultaneously: mPAP≥25mmHg, and PVR > 3 Wood units(in children PVRi > 3 WU x m2), and PAWP≤15 mmHg at rest;
* Patients diagnosed with group 1,2,4,5 PH according to the WHO classification, detailed description is as follows: Pulmonary arterial hypertension, Lung disease / chronic hypoxia associated pulmonary hypertension, Pulmonary hypertension associated with pulmonary artery stenosis / obstruction and Pulmonary hypertension caused by other multiple factors
* Take at least one pulmonary hypertension targeted drug or calcium antagonist;
* Signed written informed consent.

Exclusion Criteria:

* Patients diagnosed with pulmonary hypertension related to left heart disease;

Ages: 3 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients or inpatients with pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse drug events | through study completion, an average of 6 months
All-cause Mortality | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, M.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No